CLINICAL TRIAL: NCT02240966
Title: Symptoms and Clinical Signs of Hypogonadism in Testicular Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mikkel Bandak, MD, Rigshospitalet, Denmark
Other Study IDs: H-3-2013-1 75
Record Dates: First submitted 2014-09-08; First posted 2014-09-16 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Syndrome; Hypogonadism; Cardio-vascular Disease
Keywords: Testicular Neoplasms; Hypogonadism; Metabolic Syndrome; Treatment related late effects
MeSH Terms: conditions — Metabolic Syndrome; Hypogonadism; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the prevalence of signs and symptoms of hypogonadism in three groups of testicular cancer survivors.

DETAILED DESCRIPTION:
Recent studies have shown that metabolic syndrome is common among testicular cancer. Patients with low levels of testosterone appear to be at higher risk of metabolic syndrome.

A substantial number of testicular cancer survivors might be in a state of "compensated hypogonadism" with testosterone levels low in the normal range due to an increased LH-drive from the pituitary gland.

Whether this specific groups of testicular cancer survivors are at increased risk of cardio-vascular disease and might benefit from testosterone substitution is yet to be clarified.

ELIGIBILITY:
Inclusion Criteria:

* Earlier treatment of testicular germ cell cancer
* No sign of relapse > 1 year since latest treatment
* Testosterone < 12 nmol/L and luteinizing hormone > 8 IE/L OR
* Testosterone > 12 nmol/L and LH > 8 IE/L OR
* Testosterone and LH within their normal ranges

Exclusion Criteria:

* Testosterone substitution

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Testicular cancer survivors
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of Metabolic Syndrome in the three groups of testicular cancer survivors according to International Diabetes Federation Guidelines and US National Cholesterol Education Program Adult Treatment Panel III criteria | Up to 12 months

SECONDARY OUTCOMES:
Lean body mass (Kilogram) | Up to 12 months
  Lean body mass assessed by DXA-scan
Bone Mineral Density (Gram/cm2) | Up to 12 months
  Bone mineral density assessed by DXA-scan
Pulmonary Function: Total lung capacity, Forced vital capacity, FEV1, Diffusing capacity or of the lung for carbon monoxide | Up to 12 months
Renal function (Glomerular Filtration Rate ml/min) | Up to 12 months
  Renal function is assessed with 51Cr-EDTA
Fasting Blood Glucose | Up to 12 months
plasma-insulin | Up to 12 months
Adiponectin and leptin | Up to 12 months
Ultrasonic appearance and size of the remaining testicle | Up to 12 months
  Ultrasonic appearance and size of the remaining of testicle assessed by ultrasound
Quality of life | Up to 12 months
  Quality of Life is assessed by the EORTC QLQ-30 Questionnaire
Anxiety and depression | Up to 12 months
  Anxiety and depression is assessed by the questionnaire: Hospital Anxiety and Depression Scale (HADS)
Fatigue | Up to 12 months
  Fatigue is assessed by the questionnaire: Multidimensional Fatigue Inventory (MFI-20)

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, DMSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Bandak M, Jorgensen N, Juul A, Lauritsen J, Oturai PS, Mortensen J, Hojman P, Helge JW, Daugaard G. Leydig cell dysfunction, systemic inflammation and metabolic syndrome in long-term testicular cancer survivors. Eur J Cancer. 2017 Oct;84:9-17. doi: 10.1016/j.ejca.2017.07.006. Epub 2017 Jul 31. PMID 28772110
- [Derived] Bandak M, Jorgensen N, Juul A, Lauritsen J, Kier MGG, Mortensen MS, Oturai PS, Mortensen J, Hojman P, Helge JW, Daugaard G. Reproductive hormones and metabolic syndrome in 24 testicular cancer survivors and their biological brothers. Andrology. 2017 Jul;5(4):718-724. doi: 10.1111/andr.12355. Epub 2017 Jun 9. PMID 28598554